CLINICAL TRIAL: NCT05273554
Title: A Pilot Study to Assess Changes in Tumor Biology Following Second-line Treatment With Pembrolizumab Plus Lenvatinib in Patients With Advanced Pancreatic Ductal Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: STRATEGIC ALLIANCE: Merck (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0274; NCI-2022-02033 (Other: NCI-CTRP-Clinical Trial Reporting Process)
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Tumor; Adenocarcinoma
MeSH Terms: conditions — Neoplasms; Adenocarcinoma | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): by vein over about 30 minutes on Day 1 of each cycle.
  Interventions: Drug: Pembrolizumab; Drug: lenvatinib
- Lenvatinib (Experimental): 2 lenvatinib capsules at the same time by mouth every day while on study.
  Interventions: Drug: Pembrolizumab; Drug: lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab — Given by IV
  Other Names: KEYTRUDA®
Drug: lenvatinib — Given by PO

SUMMARY:
This is a clinical research study to learn if pembrolizumab in combination with lenvatinib can help to control pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
Primary Efficacy Objective

Corresponding Endpoint To obtain a preliminary estimate of the ORR* of the combination of pembrolizumab and lenvatinib in patients with advanced pancreatic ductal adenocarcinoma ORR, defined by the proportion of participants who have a CR or PR as determined by RECIST version

Secondary Objective

Corresponding Endpoints

• Determine progression free survival (PFS) according to RECIST version 1.1 and iRECIST.

PFS defined as the time from enrollment to the first occurrence of disease progression or death from any cause, whichever occurs first

* To estimate DOR according to RECIST v1.1 and iRECIST.
* DOR defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first
* To estimate DCR using RECIST 1.1 and with confirmatory assessment as required by iRECIST at any time during the trial.
* DCR defined as the proportion of subjects who have a CR, PR, or SD
* To evaluate the efficacy, toxicity and survival following treatment with pembrolizumab and lenvatinib • OS defined as the time from the date of enrollment to the date of death due to any cause.
* Occurrence and severity of AEs, with severity determined according to NCI CTCAE,

Exploratory Objective

Corresponding Endpoints To identify molecular (genomic, metabolic, and/or proteomic) biomarkers that may be indicative of clinical response/resistance, safety, pharmacodynamic activity, and/or the mechanism of action of pembrolizumab and lenvatinib Molecular (genomic, metabolic and/or proteomic) determinants of response or resistance to treatments, using blood and/or tumor tissue

* Change in T-cell composition of tumor as identified by multiplex immunofluorescent assay of serial biopsies obtained from patients. Tumor infiltrate will be assessed for any change in response to this therapeutic approach.
* Additional measurements will include changes in immune composition of tumor stroma, T-cell receptor composition in infiltrating T cells, and serum cytokines. Tumor infiltrate and circulating cytokines will be assessed for change in response to these therapies.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the patient must:

1. Have histologically or cytologically confirmed diagnosis of metastatic pancreatic adenocarcinoma based on pathology report
2. Have received at least one prior regimen of therapy for metastatic disease. May have received an unlimited number of treatments in the neoadjuvant or adjuvant setting prior to the appearance of metastatic disease.
3. Be willing and able to provide written informed consent for the trial.
4. Be 18 years of age on day of signing informed consent.
5. Have measurable disease based on RECIST 1.1. Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Have documented objective radiographic progression on or after stopping treatment with first-line therapy.

   Note: the same image acquisition and processing parameters should be used throughout the study for a given patient.
7. Be willing to provide tissue from a newly obtained core- or excisional biopsy of a tumor lesion from a metastatic site. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Patients for whom newly-obtained samples cannot be provided (e.g. inaccessible or patient-safety concern) may submit an archived specimen only upon agreement from Merck. The specimen must be from a biopsy site that would be accessible for at least one subsequent biopsy after initiation on the trial.
8. Has the ability to swallow and retain oral medication.
9. Has adequately controlled BP with or without antihypertensive medications, defined as BP ≤150/90 mm Hg with no change in antihypertensive medications within 1 week prior to randomization
10. Have a performance status of 0 or 1 on the ECOG performance status scale within 5 days of starting study treatment.
11. Have a predicted life expectancy of greater than 3 months.
12. Demonstrate adequate organ function as defined in Table 2. All screening labs should be performed within 10 days of treatment initiation.
13. Male subjects are eligible to participate if they agree to the following during the intervention period and for at least 30 days after the last dose of lenvatinib

    * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
    * Must agree to use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause [Appendix 5]) as detailed below:

      * Agree to use a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse with a WOCBP who is not currently pregnant. Note: Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile-vaginal penetration.

    Please note that 30 days after lenvatinib is stopped, if the subject is on pembrolizumab only, no male contraception measures are needed.
14. A female subject is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

    * Is not a WOCBP OR
    * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis), as described in Appendix 5 during the intervention period and for at least 120 days post pembrolizumab or 30 days post lenvatinib, whichever occurs last. The investigator should evaluate the potential for contraceptive method failure (i.e., noncompliance, recently initiated) in relationship to the first dose of study intervention
    * A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study intervention.
    * If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the subject must be excluded from participation if the serum pregnancy result is positive.

      * Additional requirements for pregnancy testing during and after study intervention are located in Appendix 5.
      * The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
      * Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

1. Has pancreatic tumor other than adenocarcinoma, including: acinar cell carcinoma, pancreaticoblastoma, malignant cystic neoplasms, endocrine neoplasms, squamous cell carcinoma. Patients with vater-, periampullary duodenal-. or common bile duct malignancies are also excluded. Patients with mixed tumor types (adenocarcinoma plus other) may be included if a metastatic site has been documented as containing adenocarcinoma.
2. Is currently receiving study therapy; or has participated in a study of an investigational agent and received study therapy, herbal/complementary oral- or IV medicine, or used an investigational device within 2 weeks of the first dose of this protocol's study treatment.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Had a solid organ or hematologic transplant.
5. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
6. Had a diagnoss of an additional malignancy made within 1 year prior to first dose of study treatment with the exception of curatively treated basal-cell carcinoma of the skin, squamous-cell carcinoma of the skin, localized prostate cancer, and/or curatively resected in situ cervical- and/or breast cancers.
7. Has presence of gastrointestinal condition, eg, malabsorption, that might affect the absorption of study drug.
8. Has present or progressive accumulation of pleural, ascitic, or pericardial fluid requiring drainage or diuretic drugs within 2 weeks prior to enrollment. The participant can receive diuretic drugs as needed per the treating physician, outside of the above-mentioned conditions.
9. Has radiographically detectable (even if asymptomatic and/or previously treated) central nervous system metastases and/or carcinomatous meningitis as assessed by the investigator and with radiology review.
10. Has clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study drug
11. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy (including dialysis), or laboratory abnormality that might confound the results of this trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient, in the opinion of the treating investigator.
14. Has known psychiatric- or substance-abuse disorders that would interfere with cooperation with trial requirements.
15. Has received prior therapy with lenvatinib, an anti-PD-1, anti-PD-L1, or anti PD-L2 agent, a VEGFR2 agent, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137).
16. Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
17. Has known hepatitis B or hepatitis C
18. Has received a live or live-attenuated vaccine within 30 days of planned start of study therapy (Cycle 1, Day 1). Administration of killed vaccines are allowed.
19. Is unable to tolerate a contrast enhanced CT or MRI for staging/restaging purposes
20. Has severe hypersensitivity (≥Grade 3) to pembrolizumab, lenvatinib, or any of its excipients.
21. Has had a prior anti-cancer monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to such agents administered more than 4 weeks earlier.
22. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered small molecule agent.

    * Note: patients with ≤ Grade 2 neuropathy or alopecia are an exception to this criterion and may qualify for the study.
    * Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study therapy.
23. Has had major surgery within 3 weeks prior to first dose of study interventions. Note: Adequate wound healing after major surgery must be assessed clinically, independent of time elapsed for eligibility
24. Has preexisting ≥Grade 3 gastrointestinal or non-gastrointestinal fistula.
25. Has urine protein ≥1 g/24 hours. Note: Participants with proteinuria ≥2+ (≥100 mg/dL) on urine dipstick testing (urinalysis) will undergo 24-hour urine collection for quantitative assessment of proteinuria.
26. Has a left ventricular ejection fraction (LVEF) below the institutional (or local laboratory) normal range, as determined by multigated acquisition (MUGA) or echocardiogram (ECHO).
27. Has radiographic evidence of encasement or invasion of a major blood vessel, or of intratumoral cavitation.

    NOTE: The degree of proximity to major blood vessels should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.
28. Has prolongation of QTcF interval to >480 ms.
29. Has clinically significant cardiovascular disease within 12 months from first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability.

    Note: Medically controlled arrhythmia would be permitted.
30. Has a history of arterial thromboembolism within 12 months of start of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To obtain a preliminary estimate of the ORR* of the combination of pembrolizumab and lenvatinib in patients with advanced pancreatic ductal adenocarcinoma | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Smaglo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT05273554/ICF_000.pdf